CLINICAL TRIAL: NCT02085967
Title: A 2-Part Study to Assess Potential Metabolism-Based Drug-Drug Interactions of E2006 When Coadministered With Itraconazole, Rifampin, Midazolam, or Bupropion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-004
Record Dates: First submitted 2014-03-10; First posted 2014-03-13 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Subjects
Keywords: Healthy; Metabolism; Drug-Drug Interactions
MeSH Terms: interventions — Rifampin; Itraconazole; Midazolam; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E2006 Part A (Experimental): E2006 10-mg tablets alone and in combination with rifampin 600 mg or itraconazole 200 mg
  Interventions: Drug: rifampin 600 mg; Drug: itraconazole 200 mg; Drug: E2006
- E2006 Part B (Experimental): E2006 10-mg tablets alone and in combination with midazolam 2 mg plus bupropion 75 mg
  Interventions: Drug: midazolam 2 mg with bupropion 75 mg; Drug: E2006

INTERVENTIONS:
Drug: rifampin 600 mg
  Arms: E2006 Part A
Drug: itraconazole 200 mg
  Arms: E2006 Part A
Drug: midazolam 2 mg with bupropion 75 mg
  Arms: E2006 Part B
Drug: E2006

SUMMARY:
This study will be a single center, open-label, drug-drug interaction study in healthy male and female subjects. The study will consist of 2 parts. In Part A, the effects of steady-state dosing of a strong CYP3A inhibitor (itraconazole) or inducer (rifampin) on the pharmacokinetics of E2006 and metabolites will be assessed. Approximately 30 subjects will be sequentially assigned to 1 of 2 treatment groups to receive itraconazole or rifampin in equal numbers (approximately 15 subjects per group). The itraconazole treatment group will be fully enrolled before enrollment is initiated for the rifampin treatment group. In Part B, the effects of steady-state dosing of E2006 on the pharmacokinetics of midazolam, a substrate of CYP3A, plus bupropion, a substrate of CYP2B6, will be assessed in approximately 24 subjects. The 2 study parts can be conducted in parallel.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Healthy males or females, ages 18 to 55 years
2. Body mass index greater than 18 and less than or equal to 32 kg/m2 at Screening
3. All females must be of nonchildbearing potential
4. Males who are not abstinent or have undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use, a highly effective method of contraception
5. Are willing and able to comply with all aspects of the protocol
6. Provide written informed consent

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Any subject that has a known history of malaria or has traveled to a country with known malarial risk (ie, is designated as "high" or "moderate" risk country according to the list available at http://www.cdc.gov/malaria) within the last year
2. Subjects with a history of bowel resection, any malabsorptive disorder, severe gastroparesis, or any gastrointestinal procedure for the purpose of weight loss (including LAP-BANDTM), which would slow gastric emptying and potentially affect PK profiles of E2006
3. Subjects with a known history of clinically significant drug or food allergies
4. Subjects who experienced a weight loss or gain of greater than 10% between Screening and prior to dosing
5. Subjects who had a clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
6. Subjects with any clinically abnormal symptom or organ impairment found in medical history, symptoms or signs, vital sign measurements, electrocardiogram (ECG) findings, or laboratory test results that require medical treatment found in medical history or at screening and baseline
7. Subjects known to be positive for human immunodeficiency virus, or subjects who have positive hepatitis B or hepatitis C screening test results
8. Subjects who have a history of drug or alcohol dependency or abuse (as defined by The Diagnostic and Statistical Manual of Mental Disorders V criteria) within approximately 2 years prior to Screening, or who have a positive urine drug test results at Screening or Baseline
9. Subjects who received blood products within 4 weeks, donated blood within 8 weeks, or donated plasma within 1 week of dosing
10. Subjects who used hormonal replacement therapy within 3 months prior to dosing
11. Subjects who used any drugs, over-the-counter (OTC) medications, nutritional supplements (eg, products containing St John's wort), excessive doses of vitamins (in the opinion of the principal investigator), herbal preparations, or foods or beverages known to modulate CYP (eg, CYP3A4) or transporters within 4 weeks prior to dosing, or who are unwilling to abstain from using these during the study
12. Subjects who engaged in intense physical activity within 1 week prior to Baseline (eg, weight training)
13. Subjects who smoke or have used tobacco or nicotine-containing products within 3 months prior to dosing
14. Subjects who habitually consume more than 400-mg caffeine per day
15. Subjects who participated (received investigational product) in another clinical trial less than 1 month (or 5 elimination half-lives of the investigational product) prior to dosing or who are currently enrolled in another clinical trial
16. Subjects with a disease that may influence the outcome of the study, such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism, or subjects who have any condition that would make him or her, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason

    Restrictions on concomitant medications, food and beverages:
17. Prescription drugs are prohibited within 4 weeks of dosing and OTC medications within 2 weeks prior to dosing and until the Termination Visit
18. Smoking or use of tobacco or nicotine-containing products is prohibited within 4 weeks prior to dosing and until Termination Visit
19. Intake of caffeinated beverages or food is prohibited 72 hours prior to dosing and throughout the entire study
20. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) is prohibited within 2 weeks prior to dosing until the Termination Visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): AUC(0-t) | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Area under the concentration-time curve from zero time to time of last quantifiable concentration
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): AUC(0-inf) | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Area under the concentration-time curve from zero time extrapolated to infinite time
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): Cmax | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Maximum observed concentration

SECONDARY OUTCOMES:
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): tmax | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Time at which the highest drug concentration occurs
Pharmacokinetics of E2006: AUC(0-8h) | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Area under the concentration-time curve from time zero time to 8 hours after dosing (E2006 only)
Pharmacokinetics of E2006: AUC(0-24h) | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Area under the concentration-time curve from time zero time to 24 hours after dosing (E2006 only)
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): AUC(0-72h) | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Area under the concentration-time curve from zero time to time 72 hours after dosing
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): t1/2 | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Terminal elimination phase half-life
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): CL/F | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Apparent total clearance after extravascular administration
Pharmacokinetics of E2006 and its major metabolites, M4, M9, and M10 (Part A), and midazolam, bupropion, and the hydroxylated metabolite of bupropion (Part B): AUC(0-inf), metabolite ratio | Approximately 56 Days for Part A; Approximately 42 Days for Part B
  Ratio of S,S-hydroxybupropion to S-buproprion

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development LLC, Austin, Texas, United States